CLINICAL TRIAL: NCT04520867
Title: Expansion And Evaluation Of The University Of Colorado Strength (Striving To Reactivate Esophageal And Gastric Health) Prehabilitation Program
Brief Title: STRENGTH Expansion
Status: Withdrawn | Type: Observational
Why Stopped: PI is leaving the institution
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-0246.cc; P30CA046934 (NIH)
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Esophageal Cancer; Gastroesophageal Junction Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Qualifying Subjects: Patients seen in the EGMDC for treatment planning who are recommended to receive neoadjuvant treatment followed by surgery at UCCC Metro
  Interventions: Other: STRENGTH

INTERVENTIONS:
Other: STRENGTH — Patients with esophageal (EC) and gastroesophageal junction (GEJC) cancers who are seen in the Esophageal and Gastric Multidisciplinary Clinic (EGMDC) for treatment planning and are recommended to receive neoadjuvant therapy and plan to receive treatment at UCCC Metro will be offered enrollment into the study. Patients will complete the patient reported assessments focused on QOL and physical activity on provided tablet computers during UCCC visits at specified time points. If unable to complete assessments in person they will be e-mailed to the patient via REDCap to complete. Additional data regarding dosing of chemotherapy, radiation, nutrition and surgical outcomes will be collected.
  Other Names: STRIVING TO REACTIVATE ESOPHAGEAL AND GASTRIC HEALTH

SUMMARY:
Patients seen in the EGMDC (Esophageal and Gastric Multidisciplinary Clinic) for treatment planning who are recommended to receive neoadjuvant treatment followed by surgery at UCCC Metro will be offered enrollment into the study. Patients will complete the self-assessments outlined below on provided tablet computers during UCCC visits. If unable to complete assessments in person they will be e-mailed via REDCap Survey to the patient to complete individually.

DETAILED DESCRIPTION:
Patients with esophageal (EC) and gastroesophageal junction (GEJC) cancers who are seen in the Esophageal and Gastric Multidisciplinary Clinic (EGMDC) for treatment planning and are recommended to receive neoadjuvant therapy and plan to receive treatment at UCCC Metro will be offered enrollment into the study. Patients will complete the patient reported assessments focused on QOL and physical activity on provided tablet computers during UCCC visits at specified time points. If unable to complete assessments in person they will be e-mailed to the patient via REDCap to complete. Additional data regarding dosing of chemotherapy, radiation, nutrition and surgical outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form
2. Age ≥ 18 years
3. Receiving treatment according to the STRENGTH pathway
4. Diagnosed with esophageal(EC)/gastroesophageal junction cancer(GEJC) stage IB-IIIB
5. Planning to receive neoadjuvant treatment followed by surgery at University of Colorado Cancer Center (UCCC) Metro
6. Ability to complete surveys online via an emailed REDCap survey link if unable to complete in person

Exclusion Criteria:

1. Inability to read English and complete questionnaires independently
2. Per the investigator, unable to comply with study criteria or assessments
3. Inability to receive and complete REDCap survey online

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each year the Esophageal and Gastric Multidisciplinary Clinic (EGMDC) sees nearly 75 patients with stage IB-IIIB EC/GEJC, and about 30 of those patients are treated locally at UCCC Metro. These patients are treated according to the STEGNTH pathway, which is standard of care. Patients will be approached at their EGMDC visit to discuss inclusion in the study
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 Score | pre-treatment baseline and 6 months post-surgery
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire is a validated patient self-reported tool. It assesses nine multi-item scales: five functional scales (physical, role, cognitive, emotional and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale. There are also several single-item symptom measures. Patients self-report using a 4-point Likert scale. Raw scores are transformed to a 0-100 scale, with higher scores representing better functioning/QOL and greater symptom burden.

SECONDARY OUTCOMES:
Changes in Weight | 9 months
  Documented by dietitian
Malnutrition Scores | 9 months
  This will be assessed by the dietitian on a scale of Mild, Moderate or Severe.
Dysphagia Score | 9 months
  This will be assessed by the dietitian on a scale of Mild, Moderate or Severe.
PRO CTCAE Scores | 9 months
  The Patient Reported Outcome Common Terminology Criteria for Adverse Events will measure the significance of adverse events, by the patient's determination. A library of 78 symptomatic AEs was developed for patient self-reporting. The toxicities chosen for self-reporting include symptomatic toxicities that can be reasonably reported from the patient perspective such as pain, fatigue, nausea, and cutaneous side effects. Most symptoms are characterized based upon key attributes:
  presence/absence, frequency, severity, and/or interference with usual or daily activities. Patients assess toxicities on a 5-point Likert scale with a recall period of the past 7 days.

OTHER OUTCOMES:
Godin Exercise Leisure-time Questionnaire | From baseline thru 3 and 6 months post surgery
  The Godin-Exercise Leisure-time Questionnaire has been utilized to assess self-reported leisure time, physical activity. This short form focuses on weekly frequencies of strenuous moderate, and light activity as well as engagement in regular leisure activity long enough to work up a sweat. A total weekly leisure activity score can be calculated and categorized into one of three groups: active, moderately active, or insufficiently active. This questionnaire will be modified to assess use of group versus individualized exercise as well.In this scale, a higher scale reflects more exercise.
QLQ-OES18 | From baseline thru 3 and 6 months post surgery
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Oesophageal module is a validated assessment tool to be used for patients with esophageal cancer undergoing any single or combination of treatments including esophagectomy, chemoradiation, endoscopic palliation or palliative chemotherapy and/or radiotherapy and should be used with the QLQ-C30. The QLQ-OES18 focuses on the extent to which patient have symptoms of problems during the last week in the following areas: eating, reflux, pain, trouble swallowing saliva, choking while swallowing, dry mouth, trouble with taste, trouble with coughing, trouble talking, and dysphagia. The response format is a four-point Likert scale. Responses to the questionnaires are transformed into a 0-100 scale using EORTC guidelines.
Eastern Cooperative OnCology Group Performance Status | From baseline thru 3 and 6 months post surgery
  It describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.).
Surgical Pathologic response in relation to EORTC QLQ-C30 | 6 months post surgery
  How the patient's actual disease response, on a scale of Complete, Partial, Stable disease, or No Response to treatment, relates to their EORTC QLQ-C30 Score

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States